CLINICAL TRIAL: NCT06771882
Title: Effect of Breast Milk Olfactory Stimulation Based Intervention on Preterm Infants' Feeding Outcomes
Brief Title: Effect of Breast Milk Olfactory Stimulation
Acronym: BMOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman tawfik, assistant lecture, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: olfactory stimulation
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Preterm Infant Feeding Outcomes

STUDY DESIGN:
Intervention Model Description: The researcher obtained 5cc soaked in a 2cm×2 cm piece of sterilized gauze for every intervention administration.
  * The preterm neonates were positioned in the supine position and the head turned to one side
  * The gauze was placed near the head, 2cm away from the nose for 2 minutes before feeding to stimulate an olfactory sense of preterm neonates 3 times per day (11 am, 2 pm, and 5 pm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMOS technique (Active Comparator): The researcher obtained 5cc soaked in a 2cm×2 cm piece of sterilized gauze for every intervention administration.
  * The preterm neonates were positioned in the supine position and the head turned to one side
  * The gauze was placed near the head, 2cm away from the nose for 2 minutes before feeding to stimulate an olfactory sense of preterm neonates 3 times per day (11 am, 2 pm, and 5 pm).
  Interventions: Other: BMOS technique

INTERVENTIONS:
Other: BMOS technique — The researcher obtained 5cc soaked in a 2cm×2 cm piece of sterilized gauze for every intervention administration.
  * The preterm neonates were positioned in the supine position and the head turned to one side
  * The gauze was placed near the head, 2cm away from the nose for 2 minutes before feeding to stimulate an olfactory sense of preterm neonates 3 times per day (11 am, 2 pm, and 5 pm).

SUMMARY:
Breast milk olfactory stimulation will improve preterm infants' outcomes.

DETAILED DESCRIPTION:
The researcher will explain the aim of the study and the components of the tools to the studied nurses.

* The researcher will distribute questionnaire to studied nurses for assessing their knowledge and the researcher will observe their practices regarding breast milk olfactory stimulation for premature infants.
* The researcher will be divided preterm infant randomly into two equal groups (control and study). While intervention will be directed to study group only before feeding. Both groups will be subjected to same routine care of the NICU.
* The researcher will be used PIBB scale and neonatal behavioral responses Sheet to assess the premature infants at 1st day of admission as pre intervention after routine care as "change diaper, eye care, cord care, feeding" at morning shift at ten o'clock and one o'clock in the afternoon for study and control group (pre intervention).
* The researcher will apply breast milk olfactory stimulation technique for study group only before feeding but, both groups will be subjected to same routine care of the NICU.
* The researcher will assess the effect of used olfactory stimulation technique to study group at 5th and 6th day of admission post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant has gestational of 30 >37.
* Birth weight 1000 > 2500 gm.
* Preterm infant fed oral or gavage feeding or both of them.

Exclusion Criteria:

* Preterm infants on mechanical ventilation or complicated case

Ages: 30 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
enhance preterm infant feeding outcomes | after one week from use breast milk olfactory stimulation
  Preterm Neonates Feeding Progression by use (Preterm Infant Breast feeding Behavior Scale .Scoring system. It will be classified into three categories: Low if score (8 to 10), Moderate if score (11 to 16) and Better if score (17 to 20).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital and Maternity & Gynecological Hospital affiliated to Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data is available with co responding outers on reasonable request